CLINICAL TRIAL: NCT06267807
Title: Lymphatic Phenotype in Patients With Noonan Syndrome Without a Clinical History of Lymphatic Disease
Brief Title: Lymphatic Phenotype in Noonan Syndrome Spectrum Disorders
Acronym: LENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 114369; NL84520.091.23 (Other: Protocol ID METC)
Record Dates: First submitted 2024-01-18; First posted 2024-02-20 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-04

CONDITIONS: Lymphatic System Disorders Congenital; Lymphatic Diseases; Noonan Syndrome; Lymphatic Disease
MeSH Terms: conditions — Lymphatic Diseases; Noonan Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR lymphangiography contrast injection (Other): GBCM will be administered. Any routinely used macrocyclic GBCM can be used for MR lymphangiography, we generally use Dotarem® (Gadoteric acid- gadoterate meglumine). The dose used is the same standard dose of 0.1 mmol/kg of body weight used for routine intravenous injection. The guidelines and precautions used for intravenous injection of GBCM, should be followed for MR lymphangiography.
  Subsequently, post-contrast imaging is performed (again, this will take around 20 minutes)
  Interventions: Diagnostic Test: Dynamic contrast-enhanced lymphangiography

INTERVENTIONS:
Diagnostic Test: Dynamic contrast-enhanced lymphangiography — The subject is placed supine on a detachable MR imaging table, outside the scanning room. Both inguinal regions are prepared under sterile conditions. Using Ultrasound guidance, the thoracic duct outlet at the left venous angle is identified. Under US guidance, a small 25 gauge needle is placed at the corticomedullar junction of an inguinal lymph node on each side. The needle position is confirmed and checked that there is no extravasation at saline injection under US visualization. The subject is then transferred to the MR imaging machine. First, pre-contrast imaging is performed, this takes around 20 minutes.
  Other Names: MR lymphangiography

SUMMARY:
To get a better insight into the central conducting lymphatic system in adult volunteers with Noonan Syndrome (NS) without clinical symptoms or signs of lymphatic disease compared to NS and CardioFacioCutaan syndrome patients with severe lymphatic disease

DETAILED DESCRIPTION:
Rationale: Noonan Syndrome Spectrum Disorders (NSSDs) are caused by pathogenic variants in genes of the Ras/MAPK signaling pathway, and belong to the RASopathy.

Lymphatic disease occur in 36% of patients with Noonan Syndrome (NS) during their lifetime, with different symptoms, severity, and onset. However, it is unknown how many patients with RASopathy are exactly impaired with lymph flow disorders, since many of these patients have unrecognized symptoms and go undiagnosed. For example, patients diagnosed with primary lymphedema (which implies being without known etiologic cause) may have an anatomic or functional abnormality of the central conducting lymph system that is not diagnosed as the causative lymph flow problem. With the diagnosis being based on the symptoms and not on the underlying pathophysiological mechanism, therapy will focus on diminishing symptoms and not on healing the pathophysiological cause. To eventually improve therapeutic intervention, a better understanding of the pathophysiology is necessary, and may be found by studying the central conducting lymphatic system of patients with NS and lymphatic disease, and adult volunteers with Noonan Syndrome without lymphatic disease. Objective: To get a better insight into the central conducting lymphatic system in adult volunteers with Noonan Syndrome (NS) without clinical symptoms or signs of lymphatic disease compared to NS and CardioFacioCutaan syndrome patients with severe lymphatic disease and healthy volunteers. (ongoing study: (Lymphomics; improving the understanding the anatomy of the lymphatic system and the direction and velocity of lymph flow; approved by the Medical Ethics Committee at Radboud University Medical Center Nijmegen file number 2021-7514) Study design: A single center, prospective collection of data Study population: Adult volunteers with Noonan Syndrome without (a history of) complaints or signs of lymphatic disease. Intervention: Three questionnaires (general health, lymphatic abnormalities and general MRI safety) will be taken prior to the dynamic MR lymphangiography. In addition to standard physical examination and electronic patient file screening, for inclusion and exclusion purposes. Subsequently, the MR lymphangiography will be performed. After 24 hours, the subject will be called for a follow-up by phone. Main study parameters/endpoints: the anatomy of the central lymph vessels, the velocity and direction of lymph flow, which can be compared with reference values. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participation in this study places subjects at minimal risk. Subjects will undergo placement of a small needle in an inguinal lymph node on both sides, with very little risk of bleeding and/or infection, as with other minimal invasive procedures. The dynamic MR lymphangiography will take approximately two hours

ELIGIBILITY:
Inclusion Criteria:

* Noonan Syndrome confirmed by genetic test with a class 4 or 5 pathogenic variant according to ClinVar
* 18 years and older (no restriction for sex)
* Willing and able to have MR lymphangiography scanning in the Radboudumc
* Oral and written informed consent
* None of the exclusion criteria

Exclusion Criteria:

* unsuitable for MRI (e.g. metallic objects in the body, severe claustrophobia)

  * A history of symptoms related to lymphatic disease
  * pregnancy
  * renal insufficiency
  * liver cirrhosis
  * History of surgery related to cardiovascular disease with hemodynamic consequence
  * Other genetic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Central lymphatic system anatomy and flow descriptive parameters. | Through study completion, an average of 1 year.
  Categorical assessment of the anatomy and lymphatic flow in the central lymphatic system. Including the presence or absence of the central lymphatic vessels, edema and fluid collections.
Diameter Thoracic duct | Through study completion, an average of 1 year.
  Measurements consist of the maximal diameter of the thoracic duct, the diameter at the level of the diaphragm, and the width and length of the cisterna chyli.
Lymph flow velocity | Through study completion, an average of 1 year.
  Lymph flow velocity will be determined on the dynamic MR lymphangiography by measuring the distance of contrast movement covered over time in cm/min.

OTHER OUTCOMES:
Demographics age | Demographics will be assessed before the start of the scan
  Age (years)
Demographics gender | Demographics will be assessed before the start of the scan
  Gender
Demographics | Demographics will be assessed before the start of the scan
  body height (centimeters)
Demographics weight | Demographics will be assessed before the start of the scan
  Weight (Kg)
Demographics clinical history | Demographics will be assessed before the start of the scan also used for inclusion
  Clinical histroy of lymphatic disease trough a questionnaire with yes/no questions
Demographics genetic background | Demographics will be assessed before the start of the scan also used for inclusion purposes
  Genetic background of the participant will be assessed trough questionnaire, or if available trought the electronical patient record. Both the gene, as well as C-DNA changes will be noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
No plan